CLINICAL TRIAL: NCT04436003
Title: Evaluation of "Muscle and Articulation Chains GDS Method" Treatment for Inoperable Low Back Pain Patients - a Randomised, Controlled Pilot Trial.
Brief Title: GDS Muscle and Articulation Chain Treatment for Chronic LBP and Spinal Stenosis
Acronym: GDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital of Vestfold (Other)
Collaborators: Oslo Metropolitan University (Other)
Responsible Party: Principal Investigator, Sidsel Lombardo, Physiotherapist, The Hospital of Vestfold
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 910193
Record Dates: First submitted 2020-06-02; First posted 2020-06-17 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Low Back Pain, Recurrent; Degenerative Disc Disease
Keywords: Muscle and articulation chains GDS method; pilot RCT; Oswestry Disability Index
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Degeneration

STUDY DESIGN:
Intervention Model Description: Patients are randomized into intervention or Control Group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and outcome assessor will be masked for randomisation. It is not possible to mask the patient and treatment provider.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle and Articulation chains GDS method treatment (Experimental): Participants in the intervention Group are examined and treated according to the principles of "Muscle and Articulation Chains GDS Method". They receive GDS treatment individually, up to 8 sessions of 1 hour.
  Interventions: Behavioral: Muscle and articulation chains GDS method
- Control (treatment as usual) (No Intervention): The Control Group receives standard treatment from their RGP/ doctor. Some are prescribed physiotherapy or chiropractor treatment, or they choose their own alternatives.

INTERVENTIONS:
Behavioral: Muscle and articulation chains GDS method — A physiotherapy method adapting treatment to patient's "terrain", or psychomorphology, using chosen techniques to balance tension between muscle chains, thus optimalizing posture and mouvement.
  Other Names: Les Chaines Musculaires et Articulaires Methode GDS
  Arms: Muscle and Articulation chains GDS method treatment

SUMMARY:
Our purpose is to conduct a pilot study to evaluate GDS muscle and articulation chain treatment for inoperable spine patients with degenerative changes in the lumbar spine, compared to "standard treatment" (any other chosen treatment). The pilot study will be conducted as a randomized controlled trial (RCT) to investigate feasibility and benefit of GDS muscle and articulation chain treatment on pain, function and quality of life. The pilot study will form the basis for a later full-scale randomized study and the following research questions will be addressed:

1. To what extent were the criteria for inclusion in the study suitable?
2. How did the recruitment procedure work?
3. How did the participants experience GDS treatment?
4. To what extent were the selected outcome measures suitable at the different evaluation moments, and which outcome measure tested in this pilot study would be most suitable as primary outcome measure in a full-scale study? (user experience will be included in the evaluation)
5. How was the change in the primary outcome measure (Oswestry Disability Index)?
6. What will be the estimated time for inclusion of the required number of participants in a full-scale study? (required sample size will be based on strength calculation /saving of the outcome target chosen as primary outcome measure for full scale study) The study is a pilot study with a randomized controlled design, with follow-up after 3-4 months. Thirty patients are recruited and receive baseline examination and respond to the questionnaires before randomization. The patients receive a questionnaire by mail 3-4 months after inclusion (after the treatment is completed for intervention group ). The pilot study will be one-way blinded.

DETAILED DESCRIPTION:
Design: randomized, controlled trial with intervention and control arm. Recruitment: Patients are recruited from those relegated from GPs in Vestfold to the spine surgeons at Vestfold Hospital (SIV) for assessment of surgery. Participants who qualify for the study will be contacted by the project staff member (Sidsel Lombardo) who will provide the information about the study. Participants who are interested in participating will be assessed in terms of the study's inclusion and exclusion criteria. If these are met, the participant will be explained what the study is based on in detail, both orally and in writing (appendix in REK application). The participant is then asked if he / she is still willing to participate. They will then undergo the baseline survey, fill in the forms and then sign the consent declaration. Afterwards they are randomized to GDS treatment or standard therapy. Participants have the opportunity to quit along the way without affecting their health care and regular treatment.

Inclusion criteria

* Women and men aged between 35 to 75 years, with chronic (> 3 months) low back pain, with or without irradiation in legs.
* Degenerative changes in the lumbar spine verified on MR. Exclusion criteria
* Severe psychiatric disorder
* Comorbidity that prevents the patient from performing exercises and gradually increasing general activity when the back / leg function permits it.
* Already had surgery with fixation of the lumbar spine.
* Pregnancy
* Being in process of assessing disability insurance or economic compensation for health reasons.

Randomization procedure: After baseline survey and answered questionnaire, participants will be randomized to intervention and control group using a data generated randomization sequence at a 1: 1 ratio. Statisticians at the Musculoskeletal Health Research Group (MUSKHealth.com) at OsloMet will assist with the randomization sequence.

Blinding: In this study, one cannot blind the participants nor the treating physiotherapist for which treatment they are receiving. However, research staff who collect and process data at the 3-4 month follow-up will be blinded to who is randomized to the intervention and control groups, respectively.

Intervention: The treatment group is examined and evaluated based on the principles of the "muscle and articulation chains GDS method", and receive until 8 treatments of one hour. They meet once a week in the beginning, more seldom towards the end of treatment. The participants pay for the individual treatments, but half prize of usual physiotherapy rate. The reason is that there is no extra money in SIV Hospital to provide free treatment, and that patients today pay regular rates for the same. Participants' follow-up to the intervention will be logged by the attending physiotherapist. The same applies to apostasy.

Control: The control group receives standard treatment from their GP, possibly referred to physiotherapy, chiropractor or the treatment option they prefer.

At baseline, imaging diagnostic findings regarding degenerative findings in the spine obtained from patient records will also be included. Data on function using Oswestry list f Data collection: Background variables such as age, gender, education level, marital status, mother tongue, height and weight will only be obtained at baseline (before randomization).

The same applies to mapping the risk of chronic back pain, which will be mapped using the STarT Back screening form [12].

Imaging diagnostic regarding degenerative findings in the spine obtained from patient records will also be included.

Functional data using the Oswestry list for functional limitations [10], pain using the VAS scale [8], health-related quality of life using the EQ-5D [11], risk for chronic back pain using the StarT Back screening form [12] and work ability will be obtained before and after intervention (3-4 months). A questionnaire at 3-4 months follow-up will be sent by mail, with a stamped envelope for return. Patients who do not respond will be reminded twice.

Statistical analysis and sample size: This pilot study will also be used to make a strength calculation for a full-scale RCT. Nevertheless, if we use minimum clinical important difference (MCID) estimates in primary outcome measures as a starting point for a strength calculation, we will get the following reasoning: MCID for ODI has been found to be between 8 and 10 points on the scale from 0 to 10 [10]. Assuming an expected difference between two groups of 8 ODI points with a standard deviation (SD) of 10 and significance level of 5%, then we will have 80% strength to detect this difference with a sample of 50 people in each group. We account for 15% drop-out, ie a full-scale study will require 115 patients. If the pilot study proves to be able to expect greater differences in ODI scores between the groups, then this number could be reduced, and vice versa. For this pilot study, the aim is to include totally 30 participants for intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 35-75 years, with cronic (>3 months) LBP, may have irradiation in legs.
* Degenerative changes in the lumbar spine verified on MR.

Exclusion Criteria:

* Severe psychiatric disorder.
* Comorbidity that prevents the patient from performing exercises and gradually increasing general activity when the back /leg function gradually allows it.
* Already had surgery with fixation of lumbar spine.
* Being in process of assessing disability insurance or economic compenastion for Health reasons.
* Pregnancy

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2020-10-03 (Actual); Study Completion 2020-10-03 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | 4 months
  Measures activity limitations

SECONDARY OUTCOMES:
Visual analogue scale (VAS) | 4 months
  Measures pain on a line 0-100
EQ-5D-5L | 4 months
  Health-related quality of life measurement tool
The Keele Start Back screening tool | 4 months
  Psychosocial screening profile measurement tool

CONTACTS AND LOCATIONS:
Overall Officials: Margreth Grotle, PhD, Principal Investigator — Oslo Metropolitan University
Locations (1):
- Vestfold Hospital, Larvik, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Diaz Arribas MJ, Ramos Sanchez M, Pardo Hervas P, Lopez Chicharro J, Angulo Carrere T, Ortega Molina P, Astasio Arbiza P. Effectiveness of the physical therapy Godelive Denys-Struyf method for nonspecific low back pain: primary care randomized control trial. Spine (Phila Pa 1976). 2009 Jul 1;34(15):1529-38. doi: 10.1097/BRS.0b013e3181aa2771. PMID 19564761
- See also: home page of author of books about the method — http://www.philippe-campignion.com
- See also: association for practitioners — http://www.apgds.com